CLINICAL TRIAL: NCT06672705
Title: Phase Ib Study to Assess the Efficacy and Safety of Epcoritamab in Relapsed or Refractory Post-Transplant Lymphoproliferative Disorder
Brief Title: Epcoritamab for the Treatment of Relapsed or Refractory Post Transplant Lymphoproliferative Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy Voorhees (Other)
Collaborators: AbbVie (Industry); Genmab (Industry)
Responsible Party: Sponsor-Investigator, Timothy Voorhees, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23408; NCI-2024-08887 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-Cell Lymphoma Post-Transplant Lymphoproliferative Disorder; EBV-Related Post-Transplant Lymphoproliferative Disorder; Recurrent Monomorphic Post-Transplant Lymphoproliferative Disorder; Recurrent Polymorphic Post-Transplant Lymphoproliferative Disorder; Refractory Monomorphic Post-Transplant Lymphoproliferative Disorder; Refractory Polymorphic Post-Transplant Lymphoproliferative Disorder
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (epcoritamab) (Experimental): Patients receive epcoritamab SC on days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 4-9, and day 1 of each subsequent cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR may continue to receive epcoritamab if disease progression occurs within 6 months. Patients with PR or SD continue to receive epcoritamab in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT and blood sample collection throughout the study and may undergo biopsy during screening.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Epcoritamab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013; Tepkinly
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase Ib trial tests the safety and effectiveness of epcoritamab in treating patients with post-transplant lymphoproliferative disorder (PTLD) that has come back after a period of improvement (relapsed) or has not responded to previous treatment (refractory). Epcoritamab, a bispecific antibody, binds to a protein called CD3, which is found on T cells (a type of white blood cell). It also binds to a protein called CD20, which is found on B cells (another type of white blood cell) and some lymphoma cells. This may help the immune system kill cancer cells. Giving epcoritamab may be safe and effective in treating patients with relapsed or refractory B-cell PTLD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety of treatment with epcoritamab in subjects with PTLD.

SECONDARY OBJECTIVES:

I. To estimate the Objective Response Rate (ORR), defined as the clinical response (complete response [CR] + partial response [PR]) after 3 cycles of epcoritamab.

II. To estimate the clinical benefit rate (CBR) in subjects with PTLD treated with epcoritamab.

III. To estimate the best objective response rate (BOR) in subjects with PTLD treated with epcoritamab.

IV. To estimate the progression free survival (PFS) in subjects with PTLD treated with epcoritamab.

V. To estimate the duration of complete response (DoCR) in subjects with PTLD treated with epcoritamab.

VI. To estimate the overall survival (OS) in subjects with PTLD treated with epcoritamab.

EXPLORATORY OBJECTIVES:

I. To characterize the peripheral immunophenotype changes through the course of treatment with epcoritamab in subjects with PTLD.

II. To describe the relationship of tumor microenvironment characteristics with clinical response to epcoritamab in subjects with PTLD.

III. To characterize Epstein-Barr virus (EBV) methylation alterations in EBV positive PTLDs treated with epcoritamab IV. To describe the relationship between metabolic tumor volume and response to epcoritamab in subjects with PTLD.

OUTLINE: This is a dose-escalation study of epcoritamab followed by a dose-expansion study.

Patients receive epcoritamab subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 4-9, and day 1 of each subsequent cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR may continue to receive epcoritamab if disease progression occurs within 6 months. Patients with PR or stable disease (SD) continue to receive epcoritamab in the absence of disease progression or unacceptable toxicity. Patients also undergo positron emission tomography (PET)/computed tomography (CT) and blood sample collection throughout the study and may undergo biopsy during screening.

After completion of study treatment, patients are followed up at 28 days and then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information to the sponsor, sites, and relevant study organizations.
* Age ≥ 18 years at the time of consent.
* Karnofsky scale ≥ 50% or Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Histological evidence of B-cell PTLD (any histologic subtype) following solid organ transplantation; expresses CD20; with or without EBV association.
* Treatment failure of immunosuppression reduction (ISR). NOTE: if ISR was deemed not feasible by treating physician, ISR treatment failure may be waived.
* Treatment failure of rituximab or rituximab plus any concurrent or sequentially administered chemotherapy regimen.
* Measurable disease of > 1.5 cm in diameter and/or bone marrow involvement.
* Subjects having undergone heart, lung, liver, kidney, pancreas, small intestine transplantation or a combination of the organ transplantations mentioned.
* HIV infection is allowed if viral load is undetectable at time of enrollment, CD4+ count > 200 cells/uL, and subject remains on anti-viral therapy.
* Resolution of toxicities from prior therapy to a grade that does not contraindicate trial participation in the opinion of the investigator.
* Expected survival greater than 60 days.
* Absolute neutrophil count 1.0 ≥ x 10^9/L.
* Platelets 50 ≥ x 10^9/L.
* Creatinine clearance (mL/min) ≥ 30 mL/min - Cockcroft-Gault Equation.

  * Note: Hematology and other lab parameters that are ≤ grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy.
* Bilirubin ≤ 3.0 x upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level > 3.0 mg/dL if their conjugated bilirubin is ≤ 3.0 × ULN).

  * Note: Hematology and other lab parameters that are ≤ grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy.
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN.

  * Note: Hematology and other lab parameters that are ≤ grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy.
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN.

  * Note: Hematology and other lab parameters that are ≤ grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy.
* Females of childbearing potential must have a negative serum pregnancy test within 3 days prior to registration. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided.
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 12 months after treatment the last dose of epcoritamab. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device.
* Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 12 months after the last dose of epcoritamab.
* Subjects with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the experimental regimen are eligible for the trial.
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.

Exclusion Criteria:

* Uncontrolled active (symptomatic) infection. Patients requiring systemic therapy are eligible if the infection is deemed controlled by the investigator.
* Post-transplant lymphoproliferative disorder following stem cell transplantation for hematologic malignancies or nonmalignant conditions.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study and lactating females must agree to not breastfeed while taking study drug).
* Subjects with central nervous system (CNS) involvement by PTLD.
* Seizure disorder requiring therapy (such as steroids or anti-epileptics).
* Uncontrolled concomitant illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association (NYHA) Class III or IV), unstable angina pectoris, myocardial infarction within 1 month prior to enrollment, uncontrolled cardiac arrhythmias, uncontrolled seizures, or severe non-compensated hypertension (systolic blood pressure > 180mmHg or diastolic blood pressure > 120mmHg).
* History of progressive multifocal leukoencephalopathy.
* Active Hepatitis B infection or Hepatitis C infection with positive viral polymerase chain reaction (PCR) from the blood. Subjects with active Hepatitis B infection and undetectable viral PCR from the blood will be allowed with concurrent use of entecavir suppression. Subjects with history of Hepatitis C infection (undetectable viral PCR) are allowed.
* Electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant.
* Any condition, including the presence of laboratory values which is deemed by the clinician to place the subject at an unacceptable risk or confounds the ability to interpret the data from this study.
* Live virus vaccines must not be administered within 28 days of the start of study treatment.
* Any investigational treatments must have been completed at least 4 weeks or 5 half-lives, whichever is shorter, prior to the start of study treatment. Investigational antibody therapies are not included in this requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the last dose of the study drug
  Will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) grading for cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS). The dose limiting toxicity period will be the first 28 days after the first dose of epcoritamab.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to completion of cycle 3 (1 cycle = 28 days)
  Will be defined as the number of patients who achieve complete response (CR) + partial response (PR) divided by the number of evaluable patients, and presented with the 95% binomial confidence interval. Will be assessed using Lugano (with LYRIC modification) response criteria.
Clinical benefit rate (CBR) | Up to 6 cycles (1 cycle = 28 days)
  Will be defined as clinical response (CR + PR + stable disease) after 6 cycles of epcoritamab using Lugano (with LYRIC modification) response criteria. CBR rate will be estimated and 95% confidence interval computed.
Best Overall Response Rate (ORR) | Up to 3 years
  Will be defined as the number of patients who achieve best ORR (CR + PR) at any time after treatment with epcoritamab. Will be estimated with the 95% binomial confidence interval. Will be assessed using Lugano (with LYRIC modification) response criteria.
Progression free survival | From the date of treatment initiation to date of progression or death, whichever occurs first, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method. Will be assessed using the LYRIC response criteria.
Duration of complete response | From treatment response to date of progression or death, whichever occurs first, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method. Will be assessed using the LYRIC response criteria.
Overall survival | From date of treatment initiation to date of death due to all causes, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Voorhees, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Washington University, St Louis, Missouri
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu